CLINICAL TRIAL: NCT04217460
Title: Intervention for Fluency Difficulty
Acronym: FIST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Responsible Party: Principal Investigator, Peter Howell, Professor, University College, London
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: phowell
Record Dates: First submitted 2019-12-29; First posted 2020-01-03 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2020-01

CONDITIONS: Word Finding Difficulty; Communication Disorders
MeSH Terms: conditions — Anomia; Communication Disorders | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Children screened for word-finding difficulty. Children at risk are matched with controls who do not have word-finding difficulty. Blind intervention.
Who Masked: Participant, Care Provider, Investigator
Masking Description: All details pseudo-anonymized before analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention for fluency difficulty (controls) (Active Comparator): Behavioural intervention (children practice speaking specially constructed non-word materials). Intervention is the same for both arms, here this is for controls.
  Interventions: Behavioral: Intervention for fluency difficulty
- Intervention for fluency difficulty (experimental) (Experimental): Behavioural intervention (children practice speaking specially constructed non-word materials). Intervention is the same for both arms, here this is for experimental group
  Interventions: Behavioral: Intervention for fluency difficulty

INTERVENTIONS:
Behavioral: Intervention for fluency difficulty — Children are required to speak materials they hear on recordings. The materials are not words, but contain sound sequences that occur in their language and English.

SUMMARY:
The focus of the study is to identify children with word-finding difficulty and other speech and communication difficulties such as stuttering, a procedure referred to as screening. Ideally, investigators want to screen all children in the reception classes in the schools with which investigators work. The procedures were designed so that they work with children who speak English or those whose first language is not English. A second aim concerns what teachers can do when a child does not pass the screen. Investigators have developed a type of treatment designed for children who have either word-finding difficulty or fluency difficulty. This project concerns the intervention for children with word-finding difficulty.

The treatment is conducted in a quiet room with pairs of children. The children with word-finding difficulty in each group are assessed individually for about 10 min before the treatment starts to establish a baseline for assessing improvement using a standardized task that tests for word-finding difficulty. A recording is taken, similar to that investigators obtained at the screening phase. The training takes place over three weeks (one session a week of 20-30 minutes' duration). Word-finding difficulty and fluency are reassessed at the end of the three-week period and at follow-up one week later.

DETAILED DESCRIPTION:
The focus of the study is to identify children with word-finding difficulty and other speech and communication difficulties such as stuttering, a procedure referred to as screening. Ideally, investigators want to screen all children in the reception classes in the schools with which investigators work. The procedures were designed so that they work with children who speak English or those whose first language is not English. A second aim concerns what teachers can do when a child does not pass the screen. Investigators have developed a type of treatment designed for children who have either word-finding difficulty or fluency difficulty. This project concerns the intervention for children with word-finding difficulty.

The researcher will visit every participating child at school for approximately 10 minutes. Prior to that, the researcher will speak to the child's teacher to ensure that the sessions do not clash with any important class activities. Each child will be seen individually and will listen to a number of "nonsense" words one by one and will be asked to repeat the word. The child will be told that these are funny sounding made up word. The child will be audio-recorded while speaking to the researcher.

Each audio recording is then analysed anonymously at UCL for signs of fluency or word finding difficulty. All children occasionally show these signs and they are not usually a cause of concern. Some parents are then invited to volunteer their child for the experimental word-finding training based on these results. This does not necessarily mean that they have word-finding problems (e.g. for children acting as controls). Separate information sheets indicating what this involves will be given to parents.

Parents will also be given a link to a brief online questionnaire about the child's language history that they can fill out at their own time on their phone or computer. No identifiable information are collected and every parent will be assigned a number that matches the child's participation number. Only the researchers will have access to the questionnaire. There is no obligation on parents who have been contacted to have their children participate in the training.

ELIGIBILITY:
Inclusion Criteria:

* matched to children with word-finding difficulty by age, gender and native language

Exclusion Criteria:

* none

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2018-08-24 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Non-word Repetition (NWR) | 3 weeks intervention
  This will be obtained to identify reception class children who have word finding difficulty (WFD) and fluency problems in schools. Samples of speech will be obtained to confirm children who have WFD or fluency difficulty.
Phonological Training | 3 weeks intervention
  The training procedure is delivered in a game form so that students can engage with and enjoy the test. All the following tests are conducted before and after training. Conversational speech samples are collected and analysed using a test for WFD (German, 1994) and one for fluency difficulty (Riley, 1994). Speech comprehension and letter sound knowledge tasks to assess educational impact.
Working Memory (WM) training | 3 weeks intervention
  This will involve three groups of children. For children with fluency difficulty, speech samples of about 10 minutes will be recorded before and at the end of WM training. Each speech sample will be assessed for %Stuttered Syllables (%SS) and Whole Word Repetition (%WWR) to obtain baseline measures and measurements following the intervention as well as in a follow up session. The intervention will be delivered to pairs of children. Two other groups of children who do not have fluency difficulty will take part either in a non-WM activity (group 1) using the same materials that will be used for the intervention group or the WM intervention (group 2).

CONTACTS AND LOCATIONS:
Locations (1):
- Peter Howell, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Pseudoanonymized in parents agree